CLINICAL TRIAL: NCT05060393
Title: Efficacy of Mindfulness-based Mobile Application Use in Patients With Depressive Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Basel (Other)
Responsible Party: Principal Investigator, Jan Sarlon, Principal Investigator, University of Basel
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202100452
Record Dates: First submitted 2021-09-08; First posted 2021-09-29 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Mindfulness-Based Cognitive Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Daily use of mindfulness-based mobile application for 30 days.
  Interventions: Behavioral: Mindfulness-based cognitive therapy
- Control group (No Intervention): Treatment as usual

INTERVENTIONS:
Behavioral: Mindfulness-based cognitive therapy — Mobile application, mindfulness-based therapy
  Arms: Intervention group

SUMMARY:
The presented randomized-controled study aim to assess the use of internet-based mindfulness intervention via mobile application for 30 days in patients with Major Depressive Disorder (MDD)

DETAILED DESCRIPTION:
Mindfulness-based interventions (MBI) proved to be effective in relapse prevention in MDD. Next, MBI in form of free mobile applications can be an effective augmentation of the treatment as usual (TAU) and can fill a gap in the ambulatory care. Given this background, the aim of this randomized controlled study is to assess the effectiveness of additional MBI via mobile app on the symptom severity and stress levels, compared to TAU.

ELIGIBILITY:
Inclusion Criteria:

* Depression, current ill

Exclusion Criteria:

* acute alcohol- and drug dependency, schizophrenia or psychotic disorder, severe somatic illnes, not having smartphone or not willing to use mobile application

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-10-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline self reported Depression Severity | 30 days
  Beck Depression Inventory
Change from Baseline Depression Severity | 30 days
  Hamilton Depression Rating Scale

SECONDARY OUTCOMES:
Change from baseline heart rate | 30 days
  Change in resting heart rate
Change from baseline blood pressure | 30 days
  Change in systolic blood pressure
Change from baseline respiratory rate | 30 days
  Change in resting respiratory rate
Change from baseline tobacco consumption | 30 days
  Change in daily tobacco consumption
Change from baseline alcohol consumption | 30 days
  Change in weekly alcohol consumption
Change in consumption of anxiolytics | 30 days
  Change in daily use of anxiolytic drugs

CONTACTS AND LOCATIONS:
Overall Officials: Jan Sarlon, Principal Investigator — University of Basel
Locations (1):
- Jan Sarlon, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial will be shared, after deidentification.
Supporting Information: Study Protocol, ICF
Time Frame: Immediately following publication and ending 5 years following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal.

REFERENCES:
- [Derived] Sarlon J, Doll JPK, Schmassmann A, Brand S, Ferreira N, Muehlhauser M, Urech-Meyer S, Schweinfurth N, Lang UE, Bruehl AB. Effectiveness of a Mindfulness-Based Mobile Application for the Treatment of Depression in Ambulatory Care: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2022 Mar 31;11(3):e33423. doi: 10.2196/33423. PMID 35357325